CLINICAL TRIAL: NCT01466829
Title: Clinical Effects of Parathyroid Hormone as Adjuvant Therapy for Bone Healing After Sternotomy.
Brief Title: Treatment With PTH After Sternotomy in Cardiac Surgery Patients
Acronym: PAATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Takeda (Industry); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011/386; 2011-004465-32 (EudraCT Number)
Record Dates: First submitted 2011-10-24; First posted 2011-11-08 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-08

CONDITIONS: Disruption or Dehiscence of Closure of Sternum or Sternotomy
Keywords: sternotomy; parathyroid hormone; bone healing
MeSH Terms: interventions — Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control patients treated with placebo.
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Daily injection with Parathyroid hormone
  Interventions: Drug: Parathyroid hormone

INTERVENTIONS:
Drug: Parathyroid hormone — 100 microgram daily. S.c
  Other Names: Preotact®
  Arms: Intervention
Drug: Placebo — Placebo; saline injection.
  Arms: Control

SUMMARY:
The aims of this study is to compare healing time and quality of newly formed bone in cardiac surgery patients treated with PTH post-surgically and a control group treated with saline.

DETAILED DESCRIPTION:
Heart surgery is most commonly performed through a central division of the sternum, a sternotomy. This procedure provides full overview of the thoracic cavity and access to the organs within. At the department of Cardiothoracic & Vascular Surgery at Skejby Hospital alone, over 1000 sternotomies are performed each year. When closing the sternum, the normal procedure is to use steel wires to hold the two sternal halves together. The patient receives no additional medical treatment to improve bone healing. Following surgery, sufficient healing of the sternum is important to prevent complications and to ensure a high level of life-quality for the patient. It has been shown that forces, equally to those produced during a normal cough, can displace the wire-fixated sternum by more than 2 mm. Reduced stability of the sternum has a negative impact on the healing process and increases the risk of infections. Another known complication to sternotomy is pseudoarthrosis (nonunion), which is caused by insufficient healing of the sternum and may result in instability, chronic pain and reduced quality of life. These complications result in prolonged admittance time, increased mortality and morbidity and from a financial point of view, increased treatment-costs for each patient.

Parathyroid hormone (PTH) is a well known anabolic drug and has been used to treat osteoporosis in post-menopausal women with great effect. A continuous high level of PTH decreases bone density and induces hypercalcemia, but if given once daily PTH has an anabolic effect on bone. It is being investigated if it is possible to use PTH in the treatment of other conditions, for example in the treatment of bone fractures.

Several studies, both clinical and experimental, show that PTH advances healing time and increases the quality of newly formed bone. It has also been shown to enable healing in sternal nonunion in one case-study. A recent human study of 102 osteoporotic women, with fractures of their radial bone, showed that daily injection with 20µg of the PTH-analog PTH1-34 (Teriparatide) reduces the fracture healing time. The effect of PTH on bone healing in sternum after a sternotomy has not previously been investigated.

In this study, we aim to investigate the effect of PTH on sternal healing in a clinical setup.

ELIGIBILITY:
Inclusion Criteria:

* Full sternotomy
* Not in chronic, systemic corticosteroid treatment.
* No Plavix treatment 5 days prior to surgery
* No known bone metabolic diseases.
* Replete vitamin D status (plasma 25-hydroxyvitamin D >50 nmol/l)
* Normal serum levels of Calcium, Phosphate, inorganic, alkaline phosphatase (within reference interval).
* No known risk of osteosarcoma.
* Ability to understand and cooperate with the planned examinations.
* Ability to speak and understand Danish.

Exclusion Criteria:

* Re-operation
* Use of bone wax during surgery
* Prior radiation therapy involving the skeleton
* Severely impaired renal function.
* Known allergic reactions to any of the compounds in the trial medication.
* Current treatment with digoxin
* Major medical or social problems that will be likely to preclude participation
* Severely impaired lever function
* Unknown raised levels of bone specific alkaline phosphatase.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Computer Tomography | 6 weeks (± 1 week), 3 months (± 2 weeks) and 6 months (± 2 weeks)
  Change in density of the fracture in the sternum at different time frames compared with baseline at 6 weeks.

SECONDARY OUTCOMES:
Questionnaires | Baseline, 6 weeks (± 1 week), 3 months (± 2 weeks), 6 months (± 2 weeks)
  Change of quality of life at different time frames compared with baseline.
Journal parameters | Baseline, 6 weeks (± 1 week), 3 months (± 2 weeks), 6 months (± 2 weeks)
  Admission time, blood tests, cross-clamp time, bypass time, time of mechanical ventilation, duration of surgery, pacingwires, type of operation, treatment with bisphosphonates, treatment with steroids, COLD, use of analgetics.

CONTACTS AND LOCATIONS:
Overall Officials: Per Nielsen, MD, Principal Investigator — Dept. of Cardiothoracic & Vascular Surgery, Aarhus University Hospital, Skejby
Locations (1):
- Dept. of Cardiothoracic & Vascular Surgery, AArhus University Hospital, Skejby, Aarhus N, Denmark